CLINICAL TRIAL: NCT01867476
Title: Adherence Monitoring For Substance Abuse Clinical Trials
Status: Completed | Type: Observational
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Creare, Inc. (Industry)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Other Study IDs: 2012.075EXP
Record Dates: First submitted 2013-01-29; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy Normals
  Interventions: Other: Automated Adherence Monitoring System

INTERVENTIONS:
Other: Automated Adherence Monitoring System

SUMMARY:
The purpose of this study is to determine the feasibility and accuracy of an automated adherence monitoring system, and to compare the variance between urine and oral fluid riboflavin levels when specimens are obtained 'as usual' and after a one-hour inter specimen interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 60
* Ability to give informed consent.
* Be willing and able to use the study-provided phone for taking and transmitting capsule photos.

Exclusion Criteria:

* Unwilling or unable to use a cell phone.
* Any medical, psychiatric, or other condition that, in the opinion of the investigator, would preclude safe, consistent, or useful participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Normals
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Variance between urine and oral fluid riboflavin levels when specimens are obtained 'as usual' and after a one-hour inter specimen interval | + 1, 2, 3, 4, 6 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: John Mendelson, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- Addiction & Pharmacology Research Lab, St. Luke's Hospital, San Francisco, California, United States